CLINICAL TRIAL: NCT00141700
Title: Rituximab Plus High-Dose Chemotherapy With Autologous Stem Cell Support for Poor-Prognosis Non-Hodgkin's Lymphoma
Brief Title: Study of Rituximab Plus High-Dose Chemotherapy Poor Prognosis Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: enrollment completed
Sponsor: University of Michigan Rogel Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2-51
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-12

CONDITIONS: Lymphoma, Non-Hodgkin's
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
This study is being conducted to determine the safety, side effects, and response to a combination of an established high-dose chemotherapy regimen, stem cell support and Rituximab (which is a form of immunotherapy).

DETAILED DESCRIPTION:
Combination chemotherapy is the standard treatment as initial therapy for aggressive NHL. Standard chemotherapy cures less than 40% of patients. High-dose chemotherapy with stem cell support (or transplant) is showing some positive results in patients with NHL that fail standard chemotherapy. The cure rate of this treatment is only about 50%.

Another treatment option called immunotherapy is being tested in lymphoma patients to see if adding immunotherapy to NHL treatments improves results. Rituximab, a form of immunotherapy, is an antibody (a type of protein) that attacks the CD20 protein found on lymphoma cell, which may result in the death of the lymphoma cell.

The study design is as follows: Patients with poor prognosis NHL receive rituximab as part of the peripheral blood progenitor cell mobilization process and as part of the preparative regimen in combination with high-dose chemotherapy. Granulocyte colony-stimulating factor (G-CSF) mobilized peripheral blood progenitor cells (PBPC) are collected and stored. After recovery from high-dose cyclophosphamide, patients are admitted to the hospital for transplant. The preparative regimen consists of rituximab, followed by high-dose chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, aggressive and/or intermediate grade and high-grade B cell NHL, CD20 positive.
* Histologic subtypes include follicular large cell, diffuse small cleaved cell, diffuse mixed small and large cell, diffuse large cell, anaplastic large cell, and mantle cell lymphomas.
* NHL must have high-intermediate or high International Prognostic Index (standard IPI) score at diagnosis. Mantle cell NHL is eligible regardless of IPI score.
* Complete or partial response to first-line therapy.
* Treated CNS or meningeal disease, using radiation therapy and/or intrathecal chemotherapy, is allowed. Patients with meningeal disease must have cytologically negative CSF at time of study entry.
* Cumulative total doxorubicin: <500 mg/m2
* Performance score 0-2
* Patients with a prior malignancy are eligible if they were treated with curative intent and have no evidence of active disease.
* Patients must not be pregnant or nursing.
* Informed Consent

Exclusion Criteria:

* pregnant or nursing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2003-03; Primary Completion 2005-03 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Assess progression-free survival after rituximab and high-dose chemotherapy with autologous PBPC support;

SECONDARY OUTCOMES:
Assess overall survival (OS) after rituximab and high-dose chemotherapy with PBPC support.
Assess safety and toxicity after rituximab and high-dose chemotherapy.
Assess CD20 recovery post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Raymond J. Hutchinson, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States